CLINICAL TRIAL: NCT01990313
Title: Neural Signatures of Tremor, Bradykinesia and Freezing in the Subthalamic Region on Parkinson's Disease and Their Acute and Long-Term Modulation by Subthalamic Deep Brain Stimulation.
Brief Title: Neural Signatures of Parkinson's Disease
Acronym: BrainRadio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Helen M. Bronte-Stewart, Dr, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25916
Record Dates: First submitted 2013-11-06; First posted 2013-11-21 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; DBS; Deep Brain Stimulation; Subthalamic Nucleus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Activa PC+S (Experimental)
  Interventions: Device: Activa PC+S

INTERVENTIONS:
Device: Activa PC+S — The Model 37604 Activa PC+S is a multiprogrammable device that can deliver therapeutic electrical stimulation and record bioelectric signals from leads implanted in the brain.
  Other Names: Model 37604

SUMMARY:
The purpose of this study is to provide objective measurements of abnormal movements of the body in correlation with neural activity of the brain and track how these change over time. This may allow for the development of objective evaluation of the neural activity causing abnormal movements, which may lead to the ability of the DBS system to stimulate the brain by sensing the abnormal neural activity that is causing abnormal movements.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of idiopathic Parkinson's disease, with bilateral symptoms at Hoehn and Yahr Stage greater than or equal to II.
* Documented improvement in motor signs on versus off dopaminergic medication, with a change in the Unified Parkinson's Disease Rating Scale motor (UPDRS III) score of >= 30% off to on medication.
* The presence of complications of medication such as wearing off signs, fluctuating responses and/or dyskinesias, and/or medication refractory tremor, and/or impairment in the quality of life on or off medication due to these factors.
* Subjects should be on stable doses of medications, which should remain unchanged until the DBS system is activated. After the DBS system is optimized (during which time the overall medication dose may be reduced to avoid discomfort and complications such as dyskinesias) the medication dose should remain unchanged, if possible, for the duration of the study.
* Treatment with carbidopa/levodopa, and with a dopamine agonist at the maximal tolerated doses as determined by a movement disorders neurologist.
* Ability and willingness to return for study visits, at the initial programming and after three, six and twelve months of DBS.
* Age > 18

Exclusion Criteria:

* Subjects with significant cognitive impairment and/or dementia as determined by a standardized neuropsychological battery.
* Subjects with clinically active depression, defined according to the Diagnostic and Statistical manual of Mental Disorders, Fourth Edition (DSM-IV) criteria and as scored on a validated depression assessment scale.
* Subjects with very advanced Parkinson's disease, Hoehn and Yahr stage 5 on medication (non-ambulatory).
* Age > 80.
* Subjects with an implanted electronic device such as a neurostimulator, cardiac pacemaker/defibrillator or medication pump.
* Subjects, who are pregnant, are capable of becoming pregnant, or who are breast feeding.
* Patients with cortical atrophy out of proportion to age or focal brain lesions that could indicate a non-idiopathic movement disorder as determined by MRI
* Subjects having a major comorbidity increasing the risk of surgery (prior stroke, severe hypertension, severe diabetes, or need for chronic anticoagulation other than aspirin).
* Subjects having any prior intracranial surgery.
* Subjects with a history of seizures.
* Subjects, who are immunocompromised.
* Subjects with an active infection.
* Subjects, who require diathermy, electroconvulsive therapy (ECT), or transcranial magnetic stimulation (TMS) to treat a chronic condition.
* Subjects, who have an inability to comply with study follow-up visits.
* Subjects, who are unable to understand or sign the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Bronte-Stewart, MD,MSE,FAAN, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

REFERENCES:
- [Background] Quinn EJ, Blumenfeld Z, Velisar A, Koop MM, Shreve LA, Trager MH, Hill BC, Kilbane C, Henderson JM, Bronte-Stewart H. Beta oscillations in freely moving Parkinson's subjects are attenuated during deep brain stimulation. Mov Disord. 2015 Nov;30(13):1750-8. doi: 10.1002/mds.26376. Epub 2015 Sep 11. PMID 26360123
- [Background] Blumenfeld Z, Koop MM, Prieto TE, Shreve LA, Velisar A, Quinn EJ, Trager MH, Bronte-Stewart H. Sixty-hertz stimulation improves bradykinesia and amplifies subthalamic low-frequency oscillations. Mov Disord. 2017 Jan;32(1):80-88. doi: 10.1002/mds.26837. Epub 2016 Nov 8. PMID 27859579
- [Result] Syrkin-Nikolau J, Koop MM, Prieto T, Anidi C, Afzal MF, Velisar A, Blumenfeld Z, Martin T, Trager M, Bronte-Stewart H. Subthalamic neural entropy is a feature of freezing of gait in freely moving people with Parkinson's disease. Neurobiol Dis. 2017 Dec;108:288-297. doi: 10.1016/j.nbd.2017.09.002. Epub 2017 Sep 7. PMID 28890315
- [Result] Trager MH, Koop MM, Velisar A, Blumenfeld Z, Nikolau JS, Quinn EJ, Martin T, Bronte-Stewart H. Subthalamic beta oscillations are attenuated after withdrawal of chronic high frequency neurostimulation in Parkinson's disease. Neurobiol Dis. 2016 Dec;96:22-30. doi: 10.1016/j.nbd.2016.08.003. Epub 2016 Aug 21. PMID 27553876

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Activa PC+S
Started | 15
Completed | 14
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Activa PC+S
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.97 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Resting State Beta Band Power Over Time
Description: We compared the beta band (13-30 Hz) power in the neural signal at the initial programming visit (baseline) and at the 12 month follow-up visit (1 year) after turning off deep brain stimulation therapy. Beta band power is normalized to average beta band power at the initial programming visit. Using a linear mixed model for repeated measures over time, regression beta coefficient was obtained to determine if beta power changed significantly between the initial programming and the 12 month follow-up visit.
Time Frame: Baseline and 1 Year
Population: 2 subjects excluded; 1 lost to follow-up, 1 had ECG artifact in neural signal
Measure: Number; unit: regression beta coefficient
Arm/Group | Activa PC+S
Number analyzed (Participants) | 13
regression beta coefficient | -0.28
Statistical Analysis 1: Comparison: Activa PC+S; Test type: Superiority; p = 0.038, Mixed Models Analysis

2. Primary Outcome: Sample Beta Entropy
Description: Sample entropy is a measure of estimated conditional predictability, calculated within a frequency range of a patient's local field potential. Freezers are subjects who have clinical history of freezing of gait symptoms and/or if the subject displayed freezing behavior pre-operatively or during the in-study gait tasks relative to non-freezers, those who have never experienced freezing of gait. We measured sample beta (13-30 Hz) entropy in subjects' local field potential. Higher values of sample entropy indicate lower estimated conditional predictability. Testing occurred over one day, at a range of approximately 1 month to 7 months post DBS device implantation.
Time Frame: 1 day
Population: 6 participants excluded; 3 due to tremor which may alter neural signal, 2 didn't have adequate amount of neural signal for analysis, 1 was lost to follow-up
Measure: Mean (Standard Deviation); unit: Sample Entropy
Arm/Group | Activa PC+S
Number analyzed (Participants) | 9
Sample Entropy
  Freezers: number analyzed (Participants) | 5
  Freezers | 0.407 (0.031)
  Non-freezers: number analyzed (Participants) | 4
  Non-freezers | 0.337 (0.062)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Activa PC+S
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No